CLINICAL TRIAL: NCT03982056
Title: "Float First": Categorising Factors Effecting Floating in Different Populations During Water Immersion.
Brief Title: Float First: An Index of Floating: Factors Affecting Floating in Different Populations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Heather Massey, Senior Lecturer, University of Portsmouth
Other Study IDs: TBA
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Floating Technique; Anthropometry; Lung Function
Keywords: Floating; Sculling; water safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main study group: Assessments performed:
  * Height
  * Mass
  * Body fat density
  * Bone density
  * Lean muscle density
  * Lung volume measurements
  * Floating technique
  * Buoyancy
  Interventions: Other: this is an observational study there are no interventions
- Validation group: Assessments performed:
  * Height
  * Mass
  * Body fat density
  * Bone density
  * Lean muscle density
  * Lung volume measurements
  * Floating technique
  * Buoyancy
  Interventions: Other: this is an observational study there are no interventions

INTERVENTIONS:
Other: this is an observational study there are no interventions — development of an index to provide appropriate information on a person's ability to float, based on Physiological and anthropometric characteristics

SUMMARY:
The study involves measurements of body composition using a DEXA scanner, lung function, buoyancy and floating technique. An understanding of the effects of physiological and anthropometric measures on an individual's ability to float may lead to the creation of a 'Floatability Score' to aid current public information. With this floatability score a set of actions that people of certain body types should adopt in water will be created, to tailor the current public safety messaging in an attempt to ensure more people are aware of how they can float in water

DETAILED DESCRIPTION:
Between 2000 and 2013 an average of 425 people in the UK drowned per annum, and a reported 100,000 people were involved in water-related emergencies involving search and rescue services. Approximately half had not intended to go into the water. Research identifies that in the first 1-3 minutes of immersion, during the "cold shock response" (CSR), there may be an increased probability of drowning fatalities. As a result of this, a theme of 'Float First' was created whereby individuals are advised to float for 1-3 minutes following immersion (by undertaking the minimum amount of activity possible to maximise the amount of air trapped in clothing layers and hence creating additional buoyancy) until the effects of the CSR have declined. However, a number of people have come forward indicating that despite the advice given, they are unable to float. This study is designed to establish the minimum activity level a person needs to stay afloat and combine this with anthropomorphic and physiological measures to develop advice for people of different shapes, sizes and body compositions.

ELIGIBILITY:
Inclusion Criteria:

* All participants who feel confident in water which they can stand up in, aged 18 years and older (18-29 years for Phase 1).
* The participant is willing and able to give informed consent for participation in the study.
* Be able to climb up and down a set of steps to access the swimming flume

Exclusion Criteria:

* Have allergies to water or chlorinated water.
* The participant is pregnant or suspects they may be pregnant.
* Not able to climb up and down a set of steps to access the swimming flume

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Accepting all adults able to give their own consent to participate, the investigators aim to recruit a mixture of participants of different body size, shape, sex and race
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Floating index | 2 minutes
  Describes the actions required to stay afloat

SECONDARY OUTCOMES:
Standing Height | with the two week study window
  Height of participant
Mass | with the two week study window - performed at the same time of day as the floating and DEXA scan measurements
  Mass of participant
Body composition | with the two week study window - performed at the same time of day as the floating and DEXA scan measurements
  a break down of the main components of the body (fat, lean tissue)
Lung function | with the two week study window - performed at the same time of day as the floating and DEXA scan measurements
  the volumes of the lungs namely, FVC, Tidal breathing, ERV and IRV
Buoyancy | with the two week study window - performed at the same time of day as the floating and DEXA scan measurements
  the buoyancy of the person floating in the water
Floating technique | 2 minutes
  The technique required to float

CONTACTS AND LOCATIONS:
Overall Officials: Heather Massey, PhD, Principal Investigator — University of Portsmouth
Locations (1):
- Heather Massey, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The participant's data will be anonymized and presented to interested parties as part of the groups' data. There are no plans to share the information which can be identifiable to a particular participant.